CLINICAL TRIAL: NCT06847386
Title: Research on the Effect of Hysteroscopic Metroplasty with Cold Scissors on Reproductive Outcome in Patients with Recurrent Implantation Failure
Brief Title: Effect of Hysteroscopic Metroplasty on Reproductive Outcome in Patients with RIF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22Y11906100
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Recurrent Implantation Failure; T-Shaped Uterus
Keywords: hysteroscopic metroplasty with cold scissiors; female infertility; recurrent implantation failure; reproductive outcome
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct Embryo Transfer (No Intervention): Patients in this group receive embryo transfer without hysteroscopy
- Hysteroscopy (Experimental): Patients in this group receive hysteroscopic examination. If T-shaped uterus is diagnosed during the operation, hysteroscopic metroplasty will be performed.
  Interventions: Procedure: Hysterocopic metroplasty

INTERVENTIONS:
Procedure: Hysterocopic metroplasty — If the uterine cavity is normal during intraoperative hysteroscopy, the operation will be finished and embryo transfer will be scheduled in 1 month after the operation; if the uterine cavity is narrowed or the uterine wall is coalesced, hysteroscopic metroplasty and IUD placement will be performed, and a second hysteroscopy with IUD retrieval will be performed after 2-month postoperative estrogen-progesterone treatment, then embryo transfer will be scheduled after 1-month estrogen-progesterone treatment.
  Arms: Hysteroscopy

SUMMARY:
In recent years with the continuous improvement of ART technology, it has brought new hope to infertile couples, however more than half of the patients still experience multiple transfer failures. Abnormalities in the structure of the uterine cavity are one of the main factors that lead to the failure of embryo implantation. Hysteroscopic metroplasty with cold scissors is an innovative technique of our team, in which micro-scissors are used in the procedure instead of the previous electric knife. Our previous study found that this technique has the effect of improving fertility outcomes in patients with T-shaped uterus.

Based on the previous study, this study is an open randomized controlled trial to include patients with more than 2 or more ART implantation failures. For the first time, cold knife hysteroscopic hysterectomy was used to treat patients with cryptic uterine stenosis in patients with repeated RIF implantation failures to assess the clinical efficacy of the technique and to investigate the effect of this technique on the pregnancy outcome of reimplantation of embryos in patients with repeated ART implantation failures. Meanwhile, this project is the first to study the diagnostic value of transvaginal 3D ultrasound/MRI for the assessment of uterine cavity status in patients with RIF, with a view to exploring the value of noninvasive imaging as an alternative to invasive hysteroscopy in the clinical management of RIF. The aim of the study is to provide a reference for early diagnosis and treatment of patients with repeated ART implantation failures, and to improve the pregnancy outcome of their reimplanted embryos.

ELIGIBILITY:
Inclusion Criteria:

* At least twice previous implantation failures
* Willing to receive further embryo transfer

Exclusion Criteria:

* Sturctural intrauterine lesions
* Severe adenomyosis
* Premature ovarian failure
* BMI > 35 kg/m^2
* Severe systemic disease or maligant tumor

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | From enrollment to the 18 months after the last embryo transfer
  Proportion of patients whose blood β-hCG test is positive after embryo transfer

SECONDARY OUTCOMES:
Biochemical pregnancy rate | From enrollment to the 18 months after the last embryo transfer
  Proportion of patients who have elevated blood β-hCG (> 25 mIU/mL) or positive urine immunopregnancy test, but ultrasound test reveal no gestational sac.
Clinical pregnancy rate | From enrollment to the 18 months after the last embryo transfer
  Proportion of patients who have fetal primitive heart tube pulsation tested with ultrasonography 4 weeks after embryo transfer.
Fetal implantation rate | From enrollment to the 18 months after the last embryo transfer
  Proportion of transfered embryos which develop into intrauterine gestational sacs.
Miscarriage rate | From enrollment to the 18 months after the last embryo transfer
  Proportion of patients with unintentional termination of intrauterine pregnancy at 28 gestational weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No